CLINICAL TRIAL: NCT07041749
Title: Comparison of the Efficacy of Microneedling Alone Versus Microneedling Coupled With Either Bleomycin or 5flourouracil in the Treatment of Plantar Warts
Brief Title: Microneedling Alone Versus Microneedling Coupled With Either Bleomycin or 5flourouracil in the Treatment of Plantar Warts
Acronym: plantar warts
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya magdi mohamed mahmoud, resident doctor at Dermatology, Venereology and Andrology department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Drugs in tt of plantar warts
Record Dates: First submitted 2025-03-20; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Warts of Foot
MeSH Terms: interventions — Bleomycin; Percutaneous Collagen Induction; Fluorouracil

STUDY DESIGN:
Intervention Model Description: The sample will be randomly assigned into three equal groups :
  * Group A (n=20); will be treated with combination of microneedling with saline.
  * GroupB (n=20);will be treated with combination of microneedling and topical bleomycin.
  * Group C (n=20);will be treated with combination of microneedling and topical 5-flurouracil .
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Placebo Comparator): (n=20); will be treated with combination of microneedling with saline.
  Interventions: Device: Microneedling alone
- Group B (Active Comparator): (n=20);will be treated with combination of microneedling and topical bleomycin.
  Interventions: Drug: Bleomycin; Device: Microneedling alone
- Group c (Active Comparator): (n=20);will be treated with combination of microneedling and topical 5-flurouracil .
  Interventions: Device: Microneedling alone; Drug: 5 fluorouracil

INTERVENTIONS:
Drug: Bleomycin — );will be treated with combination of microneedling and topical bleomycin .
  Arms: Group B
Device: Microneedling alone — ' Microneedling will be performed on each wart using dermapen supplied with 12 needles arranged in rows. Topical anesthetic cream will be applied for 60 min before the procedures. Microneedling will be performed on each wart using dermapen. The penetration depth will be adjusted at 2-mm, endpoint is pinpoint bleeding and the dermapen will be held by the hand in a vertical direction on the warts.
Drug: 5 fluorouracil — );will be treated with combination of microneedling and topical 5-flurouracil .
  Arms: Group c

SUMMARY:
To compare between the efficacy and safety of microneedling alone, microneedling with topical bleomycin and microneedling with 5-flurouracil in treatment of planter warts.

Microneedling will be performed on each wart using dermapen supplied with 12 needles arranged in rows. Topical anesthetic cream will be applied for 60 min before the procedures. Microneedling will be performed on each wart using dermapen. The penetration depth will be adjusted at 2-mm, endpoint is pinpoint bleeding and the dermapen will be held by the hand in a vertical direction on the warts.

Bleomycin is typically supplied in 15 U vials. The preparation will be diluted first with 7 mL normal saline ,double the amount taken from the vial by adding the same amount lidocaine (2%), so that the concentrations become 1 U/mL . The maximum total amount of bleomycin taken to each patient in one session will be 1 U/1 mL . Microneedling will be performed on the lesion using a microneedling pen type device with a 1-cm tip diameter at a 2-mm depth setting for 2-3 minutes until pinpoint bleebing occurs 1 mL of the prepared solution of bleomycin (1 U/1 mL) will be dropped on to the wart tissue using insulin syringe and occlusion will be applied for 3 hours.

5-FU is available in 10 mL vial: 500 mg/10 mL. Application of 5-FU solution will be done by dropping using an insulin syringe (1 mL)to help dropping of the solution on the warts surface. Then, the lesion will be occluded with a plaster for 3 h.

Sessions: Sessions will be performed every 2 weeks until complete cure or for maximum 6 sessions (total 3 month)

DETAILED DESCRIPTION:
Plantar warts are common cutaneous diseases on the sole caused by the human papillomavirus, with a high annual incidence rate of 14% . It is an extremely common problem which can be very painful and debilitating . HPV is a double-stranded DNA virus with more than 200 types being identified. The life cycle of HPV is closely associated with the proliferation and differentiation of epithelium. It often causes pain, which impairs quality of life of patients. First-choice treatments for common warts such as cryotherapy and salicylic acid have low-cure rates for plantar warts. Other treatments such as immunotherapy and intralesional bleomycin, which have compassionate use have higher cure rates.

Treatment for recalcitrant plantar warts remains a continuing challenge as the options for treatment have different levels of success.Topical medications and physical destruction of warts via cryotherapy, electrocautery, laser or photodynamic therapy are all common forms of treatment (Cureus,2023).

Bleomycin is an antibiotic derived from Streptomyces verticellus with antitumor and antiviral properties. It acts by DNA strand and leads to focal dermal necrosis, dyskeratosis and a neutrophil predominant inflammation .Bleomycin had been used since the seventies of last century for eliminating warts and despite almost six decades of use, yet reports and studies show discrepancies among cure rates that range from 0 up to 100% in certain circumstances. Blemoycin inhibits the deoxyribonucleic acid (DNA) and protein synthesis and hence can induce tissue death.

5-fluorouracil (5-FU) is an antimetabolite drug, used for several therapeutic purposes in dermatology, including premalignant and malignant lesions, keloid scars, vitiligo, and inflammatory skin diseases. Five-Fluorouracil (FU) is an antitumor agent blocks DNA synthesis by inhibition of pyrimidine and thymidine. Therefore, it inhibits cellular proliferation and replication. This action helps 5-FU to be used in the treatment of warts.

Microneedling is a fine needle that penetrates the skin to induce micro-injuries leading to production of collagen fibers and release of growth factors. Microneedling has been used as an adjuvant therapy helping a drug delivery and also used in treatment of various dermatologic diseases . Tissue injury by multiple needle punctures may induce local inflammation and a subsequent cell-mediated immune response against human papilloma virus.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

- 1. Children below 18. 2.Pregnant and lactating women. 3.Patients with any systemic disease or immunocompromised Patients or patients receiving any immunosuppressive drugs.

4. Impaired wound healing or imunosuppresion. 5.Patients who received any treatment for warts in the last month before study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — people aged 18 or above 18 years
Enrollment: 60 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the clinical response, specifically the decrease in the size of warts as measured by a ruler. | 2 years
  The response is categorized as:
  Complete response: Disappearance of the wart and return of normal skin markings.
  Partial response: 50% to 99% reduction in wart size.
  No or minimal response: 0% to 49% decrease in wart size

SECONDARY OUTCOMES:
Recurrence rate | 2 years
  The appearance of new wart lesions at the treated sites after complete remission during the three-month follow-up period is recorded as recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Rofaida Refaat Shehata, Assistant professor, Study Director — Assiut University; Amira ali abdelmotaleb, professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Yes